CLINICAL TRIAL: NCT04090476
Title: Impact of a High Intensity Community Exercise Group (BIG for Life) on Motor Function (i.e. Balance, Gait, Strength, Balance Confidence), Ability to Perform Activities of Daily Living, and Quality of Life Measures in Individuals With Parkinson's Disease.
Brief Title: BIG for Life: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Amy DeBlois, Assistant Professor, State University of New York - Upstate Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1441170
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
Keywords: community exercise group
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIG for Life Exercise Group (Experimental): This arm includes the entire cohort enrolled who will participate in the three times a week one hour community exercise group for a total of 8 weeks
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — During each of the exercise sessions the LSVT Big daily exercises will be performed along with functional tasks and gait/balance tasks. The functional tasks and gait/balance tasks will change weekly to monthly and all activities will be modified to the participant's mobility level.

SUMMARY:
This research study will aim to evaluate BIG for LIFE as a group exercise program, and determine whether three time a week exercise sessions with heart rate monitoring is beneficial to maintain or improve physical function, cognitive function, and quality of life over a period of 8 weeks (pre/post testing and 24 visits).

The specific objective of this study is to investigate the impact of this exercise group (BIG for LIFE) on motor functions (i.e. balance, gait, strength, balance confidence) and quality of life functions (sleep, depression, activities of daily living)

The investigators will test the following hypotheses:

1. that participation in this community-based exercise group will improve mobility level and balance confidence
2. that participation in this group will increase performance of activities of daily living as measured by self-assessment
3. that participation in this group will increase quality of life, cognition, sleep, or depression measures
4. that providing real time heart rate feedback in this group setting will increase the amount of time spent exercising in the target heart rate zone

DETAILED DESCRIPTION:
Study participants will complete a total of 24 exercise sessions (in person or via Zoom). At the initial session, participants will undergo screening and consent, physical assessments (10 meter walk test, 6 minute walk test, 5 Times Sit to Stand, and the Mini Bestest) and routine baseline medical assessments (Appearance, Pulses, BP) and complete self-assessments regarding balance (Activities Balance Confidence Questionnaire, ABC) and cognitive assessment with Trails A/B, quality of life (PDQ-39,PHQ-9, PDSS-2, FOG-q, and Patient-Specific Functional Scale); these assessments will be repeated at the final visit. In person assessments preferred but if unable due to health regulations they can be administered virtually. For virtual assessments the miniBESTest and 6 minute walk test will not be administered, all others can be administered virtually. Questionnaires will be mailed as well as instructions/materials for physical assessments for virtual assessments. Physical assessments will occur via zoom with help from family member or other individual. Participants will be also instructed in use of the heart rate monitor and will be instructed in importance of exercising at a moderate intensity.

During each of the exercise sessions the LSVT Big daily exercises will be performed along with functional tasks and gait/balance tasks. The functional tasks and gait/balance tasks will change weekly to monthly and all activities will be modified to the participant's mobility level. We will compare changes in assessment and questionnaire scores before and after completion of the 8-week (24 exercise sessions) intervention, anticipating that participants will either improve or not experience significant degradation of cognitive, physical or motor function, as can be observed in PD patients after completion of the exercise program.

Upon completion of the 8-week exercise program, assessments and questionnaires will be repeated, and the participants will be interviewed to gain anecdotal insight into their experience with the program. Using the rolling enrollment strategy, we will be able to accumulate data to provide interim insight into the progress on our study objectives, and to assess whether the number of subjects estimated is appropriate to achieve statistical power to support or reject our hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* People with Parkinson's disease age 18 or over, male or female will be included.

Exclusion Criteria:

* Persons under the age of 18 and those without a diagnosis of Parkinson's disease will be excluded from the study. Individuals with PD who are bed bound or wheelchair bound will be excluded. Scores of <23 on the MOCA will be excluded due to risk of cognitive impairments which may limit participation and ability to consent. Participants must be cleared for participation in the community exercise program by their physician.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Parkinson's Disease Questionnaire (PDQ-39) | Baseline and 8 weeks later (after 24 recorded exercise sessions)
  The PDQ-39 is a 39 item self-report questionnaire which assesses Parkinson's disease specific health related quality over the last month across 8 quality of life dimensions (activities of daily living, attention and working memory, cognition, communication, depression, functional mobility, quality of life, social relationships, social support). Items are answered on a 5 point ordinal scale (0=never, 1=occasionally, 2=sometimes, 3=often, 4=always) Lower scores reflect better quality of life. The sum of scores is divided by the maximum score and multiplied by 100.
Change in Patient Health Questionnaire (PHQ-9) | Baseline and 8 weeks later (after 24 recorded exercise sessions)
  Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Scores are added and divided by 27. Depression severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Change in Parkinson's Disease Sleep Scale - Version 2 (PDSS-2) | Baseline and 8 weeks later (after 24 recorded exercise sessions)
  The PDSS-2 is a 15 item self-report questionnaire specific to sleep quality for individuals with Parkinson's disease. It uses a 5 point scale (04=very often, 3=often, 2=sometimes, 1=occasionally, 0=never) Score ratings are added and lower scores correlate with better sleep quality.
Change in Freezing of Gait Questionairre (FOG-q) | Baseline and 8 weeks later (after 24 recorded exercise sessions)
  FOG-Q is a 16 item self-report measure used to asses Freezing of Gait (FOG) severity unrelated to falls in patients with Parkinson's disease. There are 6 items (4 items assess FOG severity and 2 items assess gait). Responses use a a 5-point ordinal scale from 0 (absence) to 4 (most severe). Total scores range from 0 to 24 with higher scores indicating more severe FOG.
Change in Activities-Specific Balance Confidence Scale (ABC) | Baseline and 8 weeks later (after 24 recorded exercise sessions)
  The Activities-specific Balance Confidence (ABC) Scale is a 16-item questionnaire/survey. Each item is rated from 0% (no confidence) to 100% (complete confidence) A higher score indicates more balance confidence.
Change in 5 times sit to stand | Baseline and 8 weeks later (after 24 recorded exercise sessions)
  Lower extremity strength measure
Change in 3M Backwards Walk Test | Baseline and 8 weeks later (after 24 recorded exercise sessions)
  Timed measure of Backwards Walk over the distance of 3M.
Change in 10 meter walk test | Baseline and 8 weeks later (after 24 recorded exercise sessions)
  Gait speed measure
Change in 6 minute walk test | Baseline and 8 weeks later (after 24 recorded exercise sessions)
  Walking Endurance Measure
Change in Mini-BESTest | Baseline and 8 weeks later (after 24 recorded exercise sessions)
  The Mini-BESTest is a measure of dynamic balance, functional mobility, and gait. It consists of 14 items under the sections of anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait. It is scored out of 28 points with a 3-level ordinal scale (0-2) with higher scores indicating better balance.
Change in Patient Specific Functional Scale (PSFS) | Baseline and 8 weeks later (after 24 recorded exercise sessions)
  This is a questionnaire to quantify activity limitation and measure functional outcomes. Participants choose up to 7 functional activities to rate on an 11 point ordinal scale from 0=unable to perform activity to 10= able to perform at the same level as before the problem. Total score=sum of the activity scores/number of activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Rock Steady Boxing Gym, Liverpool, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDonnell MN, Rischbieth B, Schammer TT, Seaforth C, Shaw AJ, Phillips AC. Lee Silverman Voice Treatment (LSVT)-BIG to improve motor function in people with Parkinson's disease: a systematic review and meta-analysis. Clin Rehabil. 2018 May;32(5):607-618. doi: 10.1177/0269215517734385. Epub 2017 Oct 5. PMID 28980476
- [Background] Janssens J, Malfroid K, Nyffeler T, Bohlhalter S, Vanbellingen T. Application of LSVT BIG intervention to address gait, balance, bed mobility, and dexterity in people with Parkinson disease: a case series. Phys Ther. 2014 Jul;94(7):1014-23. doi: 10.2522/ptj.20130232. Epub 2014 Feb 20. PMID 24557655
- [Background] Ebersbach G, Ebersbach A, Edler D, Kaufhold O, Kusch M, Kupsch A, Wissel J. Comparing exercise in Parkinson's disease--the Berlin LSVT(R)BIG study. Mov Disord. 2010 Sep 15;25(12):1902-8. doi: 10.1002/mds.23212. PMID 20669294
- [Background] Phannarus H, Muangpaisan W, Siritipakorn P, Chotinaiwattarakul W. Cognitive profiles and optimal cut-offs for routine cognitive tests in elderly individuals with Parkinson's disease, Parkinson's disease dementia, Alzheimer's disease, and normal cognition. Psychogeriatrics. 2020 Jan;20(1):20-27. doi: 10.1111/psyg.12451. Epub 2019 Mar 25. PMID 30912230
- [Background] Bloem BR, Marinus J, Almeida Q, Dibble L, Nieuwboer A, Post B, Ruzicka E, Goetz C, Stebbins G, Martinez-Martin P, Schrag A; Movement Disorders Society Rating Scales Committee. Measurement instruments to assess posture, gait, and balance in Parkinson's disease: Critique and recommendations. Mov Disord. 2016 Sep;31(9):1342-55. doi: 10.1002/mds.26572. Epub 2016 Mar 4. PMID 26945525
- [Background] Martinez-Martin P, Jeukens-Visser M, Lyons KE, Rodriguez-Blazquez C, Selai C, Siderowf A, Welsh M, Poewe W, Rascol O, Sampaio C, Stebbins GT, Goetz CG, Schrag A. Health-related quality-of-life scales in Parkinson's disease: critique and recommendations. Mov Disord. 2011 Nov;26(13):2371-80. doi: 10.1002/mds.23834. Epub 2011 Jul 6. PMID 21735480
- [Background] Trenkwalder C, Kohnen R, Hogl B, Metta V, Sixel-Doring F, Frauscher B, Hulsmann J, Martinez-Martin P, Chaudhuri KR. Parkinson's disease sleep scale--validation of the revised version PDSS-2. Mov Disord. 2011 Mar;26(4):644-52. doi: 10.1002/mds.23476. Epub 2011 Feb 10. PMID 21312275